CLINICAL TRIAL: NCT02709044
Title: Randomized Trial of Standard vs. Enhanced Hydration in Patients With a Diagnosis of Acute Pancreatitis Within the First Hour of the Diagnosis
Brief Title: Fluid Resuscitation in Acute Pancreatitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Vanja Giljaca, M.D. PhD, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP01
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatitis
Keywords: Acute pancreatitis; Fluid resuscitation; Crystalloids
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate

ARMS (2):
- Ringer lactate 20 mL/kg (Experimental): This group of subjects will receive a bolus of 20 ml / kg of Ringer's solution for infusion within first hour of the diagnosis
  Interventions: Drug: Ringer lactate
- Ringer lactate 40 ml/kg (Experimental): This group of subjects will receive a bolus of 40 ml / kg of Ringer's solution for infusion within first hour of the diagnosis
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Ringer lactate

SUMMARY:
The aim of this study is to establish the influence of early administration of a bolus of intravascular fluid in patients with a diagnosis of acute pancreatitis on the course and outcome of disease.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical trial of standard versus enhanced hydration in patients diagnosed with acute pancreatitis within the first hour of diagnosis.

Patients admitted in the Emergency Department with the clinical suspicion of acute pancreatitis will be processed through the history, physical examination and laboratory findings. The diagnosis of acute pancreatitis is established by the presence of 2 of the 3 following criteria: typical abdominal pain, serum amylase and / or lipase greater than three times the upper limit of normal, and characteristic findings from abdominal imaging. Patients will be informed about the study protocol and the possible risks and adverse events, after which they will be asked to accept participation in the study. Acceptance of participation will be confirmed by signed informed consent.

After acceptance patients will be randomized by computer-generated sequences of random numbers in the two groups Group one (1) will receive a bolus of fluid 20 ml / kg of Ringer's solution for infusion within one hour of the diagnosis and the group two (2) will receive a bolus of fluid 40 ml / kg of Ringer's solution for infusion within one hour of the diagnosis. All patients who have the diagnosis of acute pancreatitis, but did not agree to participate in research or have some other exclusion criteria will be treated according to the standards of good clinical practice and the recommendations of the current clinical guidelines for the treatment of acute pancreatitis. Exclusion criteria beside refusal to sign informed consent are: age less than 18 years, pregnancy, patients with physical signs of heart failure, previously known congestive heart failure (NYHA III - IV) and severe kidney disease more than one month before the diagnosis of acute pancreatitis (defined as severe reduction in eGFR less than 30 ml/min/1.73 m2). Patients who develop acute renal failure as a result of acute pancreatitis will be involved in research .

Given the importance of early hydration in patients with acute pancreatitis and the lack of clearly defined dose of administered fluid in the current literature, aim of this study was to determine the influence of the size of the dose bolus of intravascular fluid after the diagnosis of acute pancreatitis in the further course and outcome of disease.

The study will be conducted in the Emergency Department, Clinical Hospital Centre, Rijeka.

ELIGIBILITY:
Inclusion Criteria:

All patients with diagnosis of acute pancreatitis.

Exclusion Criteria:

1. Refusal to sign informed consent
2. Age less than 18 years
3. Pregnancy
4. Patients with physical signs of heart failure,
5. Previously known congestive heart failure ( NYHA III - IV )
6. Severe kidney disease more than one month before the diagnosis of acute pancreatitis (defined as severe reduction in eGFR less than 30 ml/min/1.73 m2) . Patients who develop acute renal failure as a result of acute pancreatitis will be involved in research .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of mortality | Until hospital discharge or maximum of 1 month
  Number of participants with fatal outcome during hospitalisation
Development of severe pancreatitis | Until hospital discharge or maximum of 1 month
  Number of participants with severe pancreatitis during hospitalisation (according to revised Atlanta criteria)

SECONDARY OUTCOMES:
Development of peripancreatic collection | Until hospital discharge or maximum of 1 month
  Number of participants with development of peripancreatic collection during hospitalisation
Development of pancreatic collection infection | Until hospital discharge or maximum of 1 month
  Number of participants with development of pancreatic collection infection during hospitalisation
Development of systemic inflammatory response syndrome (SIRS) | Until hospital discharge or maximum of 1 month
  Number of participants with development of systemic inflammatory response syndrome (SIRS)
Development of metabolic acidosis | Until hospital discharge or maximum of 1 month
  Number of participants with development of metabolic acidosis
Development of acute respiratory distress syndrome (ARDS ) defined according to the current Berlin definition | Until hospital discharge or maximum of 1 month
  Number of participants with development of acute respiratory distress syndrome (ARDS ) defined according to the current Berlin definition
Adverse events | Until hospital discharge or maximum of 1 month
  All events during the treatment of patients who may or may not be associated with acute pancreatitis and / or replacement of fluids

CONTACTS AND LOCATIONS:
Overall Officials: Vanja Giljača, M.D. PhD, Study Chair — University Hospital Rijeka
Locations (1):
- UHRijeka, Rijeka, Rijeka, Croatia

REFERENCES:
- [Background] Dugernier T, Starkel P, Laterre PF, Reynaert MS. Severe acute pancreatitis: pathophysiologic mechanisms underlying pancreatic necrosis and remote organ damage. Acta Gastroenterol Belg. 1996 Jul-Sep;59(3):178-85. PMID 9015927
- [Background] Cuthbertson CM, Christophi C. Disturbances of the microcirculation in acute pancreatitis. Br J Surg. 2006 May;93(5):518-30. doi: 10.1002/bjs.5316. PMID 16607683
- [Background] Zhao G, Zhang JG, Wu HS, Tao J, Qin Q, Deng SC, Liu Y, Liu L, Wang B, Tian K, Li X, Zhu S, Wang CY. Effects of different resuscitation fluid on severe acute pancreatitis. World J Gastroenterol. 2013 Apr 7;19(13):2044-52. doi: 10.3748/wjg.v19.i13.2044. PMID 23599623
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Bradley EL 3rd. A clinically based classification system for acute pancreatitis. Summary of the International Symposium on Acute Pancreatitis, Atlanta, Ga, September 11 through 13, 1992. Arch Surg. 1993 May;128(5):586-90. doi: 10.1001/archsurg.1993.01420170122019. PMID 8489394
- [Background] Vege SS, Chari ST. Organ failure as an indicator of severity of acute pancreatitis: time to revisit the Atlanta classification. Gastroenterology. 2005 Apr;128(4):1133-5. doi: 10.1053/j.gastro.2005.02.059. No abstract available. PMID 15825098
- [Background] Thoeni RF. The revised Atlanta classification of acute pancreatitis: its importance for the radiologist and its effect on treatment. Radiology. 2012 Mar;262(3):751-64. doi: 10.1148/radiol.11110947. PMID 22357880
- [Background] Vege SS, Gardner TB, Chari ST, Munukuti P, Pearson RK, Clain JE, Petersen BT, Baron TH, Farnell MB, Sarr MG. Low mortality and high morbidity in severe acute pancreatitis without organ failure: a case for revising the Atlanta classification to include "moderately severe acute pancreatitis". Am J Gastroenterol. 2009 Mar;104(3):710-5. doi: 10.1038/ajg.2008.77. Epub 2009 Feb 3. PMID 19262525
- [Background] Petrov MS, Windsor JA. Classification of the severity of acute pancreatitis: how many categories make sense? Am J Gastroenterol. 2010 Jan;105(1):74-6. doi: 10.1038/ajg.2009.597. Epub 2009 Oct 20. PMID 19844203
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Ranson JH, Rifkind KM, Roses DF, Fink SD, Eng K, Spencer FC. Prognostic signs and the role of operative management in acute pancreatitis. Surg Gynecol Obstet. 1974 Jul;139(1):69-81. No abstract available. PMID 4834279
- [Background] Blamey SL, Imrie CW, O'Neill J, Gilmour WH, Carter DC. Prognostic factors in acute pancreatitis. Gut. 1984 Dec;25(12):1340-6. doi: 10.1136/gut.25.12.1340. PMID 6510766
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Singh VK, Wu BU, Bollen TL, Repas K, Maurer R, Johannes RS, Mortele KJ, Conwell DL, Banks PA. A prospective evaluation of the bedside index for severity in acute pancreatitis score in assessing mortality and intermediate markers of severity in acute pancreatitis. Am J Gastroenterol. 2009 Apr;104(4):966-71. doi: 10.1038/ajg.2009.28. Epub 2009 Mar 17. PMID 19293787
- [Background] Balthazar EJ. Staging of acute pancreatitis. Radiol Clin North Am. 2002 Dec;40(6):1199-209. doi: 10.1016/s0033-8389(02)00047-7. PMID 12479706
- [Background] Juneja D, Gopal PB, Ravula M. Scoring systems in acute pancreatitis: which one to use in intensive care units? J Crit Care. 2010 Jun;25(2):358.e9-358.e15. doi: 10.1016/j.jcrc.2009.12.010. Epub 2010 Feb 10. PMID 20149591
- [Background] Schutte K, Malfertheiner P. Markers for predicting severity and progression of acute pancreatitis. Best Pract Res Clin Gastroenterol. 2008;22(1):75-90. doi: 10.1016/j.bpg.2007.10.013. PMID 18206814
- [Background] Wu BU, Johannes RS, Sun X, Tabak Y, Conwell DL, Banks PA. The early prediction of mortality in acute pancreatitis: a large population-based study. Gut. 2008 Dec;57(12):1698-703. doi: 10.1136/gut.2008.152702. Epub 2008 Jun 2. PMID 18519429
- [Background] Haydock MD, Mittal A, van den Heever M, Rossaak JI, Connor S, Rodgers M, Petrov MS, Windsor JA; Pancreas Network of New Zealand. National survey of fluid therapy in acute pancreatitis: current practice lacks a sound evidence base. World J Surg. 2013 Oct;37(10):2428-35. doi: 10.1007/s00268-013-2105-7. PMID 23720122
- [Background] Khajavi MR, Etezadi F, Moharari RS, Imani F, Meysamie AP, Khashayar P, Najafi A. Effects of normal saline vs. lactated ringer's during renal transplantation. Ren Fail. 2008;30(5):535-9. doi: 10.1080/08860220802064770. PMID 18569935
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Nasr JY, Papachristou GI. Early fluid resuscitation in acute pancreatitis: a lot more than just fluids. Clin Gastroenterol Hepatol. 2011 Aug;9(8):633-4. doi: 10.1016/j.cgh.2011.03.010. Epub 2011 Mar 21. No abstract available. PMID 21421079
- [Background] Warndorf MG, Kurtzman JT, Bartel MJ, Cox M, Mackenzie T, Robinson S, Burchard PR, Gordon SR, Gardner TB. Early fluid resuscitation reduces morbidity among patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):705-9. doi: 10.1016/j.cgh.2011.03.032. Epub 2011 Apr 8. PMID 21554987
- [Background] Wall I, Badalov N, Baradarian R, Iswara K, Li JJ, Tenner S. Decreased mortality in acute pancreatitis related to early aggressive hydration. Pancreas. 2011 May;40(4):547-50. doi: 10.1097/MPA.0b013e318215368d. PMID 21499208
- [Background] Stimac D, Poropat G. Rational therapy of acute pancreatitis. Dig Dis. 2010;28(2):310-6. doi: 10.1159/000319406. Epub 2010 Sep 1. PMID 20814204
- [Background] Tenner S. Initial management of acute pancreatitis: critical issues during the first 72 hours. Am J Gastroenterol. 2004 Dec;99(12):2489-94. doi: 10.1111/j.1572-0241.2004.40329.x. PMID 15571599
- [Background] Aggarwal A, Manrai M, Kochhar R. Fluid resuscitation in acute pancreatitis. World J Gastroenterol. 2014 Dec 28;20(48):18092-103. doi: 10.3748/wjg.v20.i48.18092. PMID 25561779
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) adopts Consolidated Guideline on Good Clinical Practice in the Conduct of Clinical Trials on Medicinal Products for Human Use. Int Dig Health Legis. 1997;48(2):231-4. No abstract available. PMID 11656783
- [Background] Werner J, Hartwig W, Uhl W, Muller C, Buchler MW. Useful markers for predicting severity and monitoring progression of acute pancreatitis. Pancreatology. 2003;3(2):115-27. doi: 10.1159/000070079. PMID 12748420
- [Background] Isenmann R, Runzi M, Kron M, Kahl S, Kraus D, Jung N, Maier L, Malfertheiner P, Goebell H, Beger HG; German Antibiotics in Severe Acute Pancreatitis Study Group. Prophylactic antibiotic treatment in patients with predicted severe acute pancreatitis: a placebo-controlled, double-blind trial. Gastroenterology. 2004 Apr;126(4):997-1004. doi: 10.1053/j.gastro.2003.12.050. PMID 15057739
- [Background] Banks PA, Freeman ML; Practice Parameters Committee of the American College of Gastroenterology. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006 Oct;101(10):2379-400. doi: 10.1111/j.1572-0241.2006.00856.x. No abstract available. PMID 17032204
- [Background] Khan AA, Parekh D, Cho Y, Ruiz R, Selby RR, Jabbour N, Genyk YS, Mateo R. Improved prediction of outcome in patients with severe acute pancreatitis by the APACHE II score at 48 hours after hospital admission compared with the APACHE II score at admission. Acute Physiology and Chronic Health Evaluation. Arch Surg. 2002 Oct;137(10):1136-40. doi: 10.1001/archsurg.137.10.1136. PMID 12361419